CLINICAL TRIAL: NCT02811107
Title: Evaluation of Anxiety in Surgery Preoperative Area (ASDT)
Acronym: ASDT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0075
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Preoperative Area
Keywords: anxiety; pain; preoperative area; premedication
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in preoperative area: Patients in preoperative area before surgery or interventional procedure will complete questionnaires on tablet computers
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Completion of questionnaires on tablet computers in the preoperative area by 6 nurse anesthetists, 1 hospital physician and 1 resident physician.

SUMMARY:
Anxiety is associated with discomfort but also with an increased risk of pain and/or analgesic consumption. A prescription of anxiolytics is very common in pre-anesthetic consultation but without considering the real anxiety level of the patients. The objective of this premedication is mainly to improve patient comfort, to reduce patient anxiety and to improve patient cooperation.

According to a study conducted in the 1990s, 40 to 80% of patients are anxious before surgery.

Consequences of anxiety are somatic (tachycardia, hypertension, difficulty to falling asleep), behavioural (aggressiveness, regression, fight against anaesthesia induction) and postoperative pain.

Preoperative area is a place of convergence for patients who need surgery or an interventional procedure.

Staying in the preoperative area may be a source of anxiety and may affect the patient management.

The investigators will interview patients undergoing surgery or interventional procedure to assess their level of anxiety, pain and their experiences during their stay in preoperative area. The objective is to analyse the level of anxiety and / or pain and their clinical consequences, and then to assess the relationship with any potential premedication.

ELIGIBILITY:
Inclusion Criteria:

* Patient in preoperative area before surgery or interventional procedure
* Patient to receive general anesthesia, local, locoregional, sedation,
* Agreeing to participate in the study after receiving information note,
* ≥ 18 years of age.

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in preoperative area before surgery or interventional procedure
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of anxiety in preoperative area, by using 3 questionnaires. | Day 0
  With 3 questionnaires:
  * visual analog scale of anxiety
  * APAIS score
  * COVI Score

SECONDARY OUTCOMES:
Evaluation of sedation | Day 0
  Scale of sedation (during the stay in preoperative area)
Evaluation of pain | Day 0
  visual analog scale of pain (during the stay in preoperative area)
Experiences of patient | Day 0
  questionnaire (during the stay in preoperative area)
Evaluation of patient premedication | Day 0
  questionnaire (during the stay in preoperative area)